CLINICAL TRIAL: NCT03234790
Title: A Controlled Dose-Response Human Study to Develop a Signature of Occupational Diesel Exhaust Exposure
Brief Title: Human Study to Develop a Signature of Occupational Diesel Exhaust Exposure
Acronym: DICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Government of Alberta (Other Government); Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Christopher Carlsten, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: H16-03053
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Experimental
Keywords: Diesel Exhaust; Air Pollution; Airway Responsiveness; Proteomics; Urine PAH Metabolites

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filtered Air Exposure (Active Comparator): Exposure for 4 hours to filtered air
  Interventions: Other: Filtered Air Exposure
- Diesel Exhaust Exposure (Experimental): Volunteers exposed to different concentrations of diesel exhaust
  Interventions: Other: Diesel Exhaust Exposure

INTERVENTIONS:
Other: Filtered Air Exposure — Exposure to Filtered air
  Arms: Filtered Air Exposure
Other: Diesel Exhaust Exposure — Diesel exposure to different concentrations at different times: 20, 50 and 150ug/m3
  Arms: Diesel Exhaust Exposure

SUMMARY:
Strong scientific understanding of how emissions from diesel engines impact the lungs could improve policies and regulations protecting workers exposed to diesel exhaust. Accordingly, we are recruiting healthy volunteers who are non-smokers to participate in our study. Volunteers sit in a room for four hours and breathe either clean filtered air or air that contains pollution at various concentrations similar to occupational settings such as bus and ferry terminals where diesel engines are used. A respirologist assesses the volunteer's lung health and clinical samples are taken. We are equipped with advanced molecular biology tools to measure different molecules and compare samples from our volunteer subjects following exposure to clean air or diesel exhaust. Our research aim is to find a simple, clinically relevant strategy that can be used to measure the impact of diesel exhaust on workers' lung health. This knowledge will empower regulators, companies, and ultimately workers to better manage their health risks. Our research aims to provide specific data to help regulators to make informed decisions about the risks of diesel exhaust exposure.

DETAILED DESCRIPTION:
1. Purpose: Over 100,000 employees in Alberta are inadvertently exposed to diesel exhaust at work because of wide use of diesel engines in vehicles and machines used in road construction, trucking, forestry, oil extraction and mineral mining. Although ambient air monitoring of DE exposure exists in some occupational settings, ambient air monitoring depends heavily on surrogate models and may yield a distorted picture of past exhaust exposure. Thus, a clear exposure limit based on bio-monitoring is needed to adequately protect the workers.
2. Objective: Our research aims to establish the relationship between exposure concentration and biological effect as an aid to determination of reference ranges for acceptable exposure.
3. Hypotheses and Aims:

   Hypothesis 1: Diesel exhaust (DE) inhalation elicits a characteristic protein output, in a dose-dependent manner.

   Aim 1. Demonstrate, using a proteomic analysis of serum and urine, a signature that acutely increases in response to a range of occupationally relevant DE concentrations.

   Hypothesis 2: DE inhalation increases concentrations of metabolites of polyaromatic hydrocarbons (PAH) in urine, in a dose-dependent manner.

   Aim 2. Ascertain the range of PAH metabolites accumulation in urine following acute exposure to a range of occupationally relevant DE concentrations.

   Hypothesis 3: DE inhalation alters the airway responsiveness to a contractile stimulus, in a dose-dependent manner, and that alteration is associated with changes in a combined proteomic/PAH-metabolomic signature.

   Aim 3: Determine the dose-response slope to methacholine, in response to a range of occupationally relevant DE concentrations, and correlate changes in this slope to changes in proteins and metabolites.

   Additionally, we aim to establish the relationship between a range of controlled DE exposure concentrations and sleep quality and breathing in sleep through the sub-study component.
4. Justification:

   Our work will inform decision makers and stakeholders in creating evidence-based policies to limit occupational diesel exhaust exposure based on relevant biology.
5. Research Method:

   This is an order-randomized, double-blinded, crossover human exposure study.

   This project aims to determine markers of DE exposure that can be used in an occupational setting. Therefore, we will use a range of occupational exposure levels to appropriately contextualize our results. For this, 20 healthy participants will be exposed to a control condition and 3 different levels of DE concentration, each for a period of 4 hours, in a randomized order. Each exposure will be separated by a washout period of two weeks. The levels will be DE titrated to 20, 50 and 150 ug/m3 PM2.5, and the control exposure will be filtered air (FA).

   Participants will undergo a methacholine challenge and will provide urine and blood samples before and after exposures to analyze lung function and biological responses.

   If participants consent to participation in the sleep sub-study, they will be provided with additional questionnaires throughout their visits pertaining to their sleep quality. The participants will be provided with an Alice NightOne sleep monitor and instructions on how to operate the equipment. The sleep monitor will be hooked up by the participant at home when they are about to sleep, following an exposure, and will monitor their sleep patterns for that night.
6. Statistical Analysis:

First, the changes in clinical parameters (methacholine PC20 and dose response slope) and serum blood protein abundance between pre- and post-exposure will be determined. These 'delta' values will be statistically compared across exposures using linear mixed effects models using R program, as outlined in our previous publications from similarly-designed protocols from our group. Values of p<0.05 will be considered significant throughout, with adjustments for multiple comparisons. Although the 2-week washout period is intended to minimize the likelihood of carryover effects, we will formally assess for this by including a term for order of exposures in the models.

Analyses for the sleep component will be performed at the Hospital of Ottawa and will be completed through a linear or logistic mixed effects model, as applicable using the R program. Similar methods to data collected from the main study. Data interpretation will be completed through a software algorithm on the local server.

ELIGIBILITY:
Inclusion Criteria:

1. 19-49 years
2. Non-smokers
3. No physician diagnosed asthma

Exclusion Criteria:

1. Pregnant/breastfeeding
2. Using inhaled corticosteroids
3. Co-existing medical conditions (as assessed by the primary investigator)
4. Taking part in another study that involves taking medications.
5. Abnormal lung function based on screening spirometry
6. Cardiac diagnosis or arrhythmia is discovered during the screening process

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Serum proteome in response to DE exposure | 4 hours & 24 hours
  Serum from each experimental condition will be analyzed by liquid chromatography-mass spectrometry (LC-MS/MS) to observe any changes between the baseline and listed time points

SECONDARY OUTCOMES:
Urine proteins in response to DE exposure | 4 hours & 24 hours
  Urine from each experimental condition will be analyzed by liquid mass chromatography to observe any changes between the baseline and listed time points.
Polycyclic Aromatic Hydrocarbons (PAH) metabolites in response to DE exposure | 4 hours & 24 hours
  PAH metabolites in urine samples will be analyzed by HPLC to observe any changes between the baseline and listed time points.
Sleep quality | baseline versus 24 hours post-exposure
  Sleep quality will be assessed by level 3 overnight monitor and questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carlsten, MD, MPH, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia - VGH site, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guest PC, Gottschalk MG, Bahn S. Proteomics: improving biomarker translation to modern medicine? Genome Med. 2013 Feb 27;5(2):17. doi: 10.1186/gm421. eCollection 2013. No abstract available. PMID 23445684
- [Background] Huang W, Smith TJ, Ngo L, Wang T, Chen H, Wu F, Herrick RF, Christiani DC, Ding H. Characterizing and biological monitoring of polycyclic aromatic hydrocarbons in exposures to diesel exhaust. Environ Sci Technol. 2007 Apr 15;41(8):2711-6. doi: 10.1021/es062863j. PMID 17533828
- [Background] Morgott DA. Factors and Trends Affecting the Identification of a Reliable Biomarker for Diesel Exhaust Exposure. Crit Rev Environ Sci Technol. 2014 Aug;44(16):1795-1864. doi: 10.1080/10643389.2013.790748. PMID 25170242
- [Derived] Orach J, Rider CF, Yuen ACY, Schwartz C, Mookherjee N, Carlsten C. Controlled Diesel Exhaust Exposure Induces a Concentration-dependent Increase in Airway Inflammation: A Clinical Trial. Ann Am Thorac Soc. 2023 Jun;20(6):834-842. doi: 10.1513/AnnalsATS.202209-762OC. PMID 36930796